CLINICAL TRIAL: NCT01735136
Title: Efficacy and Safety of InSan Bamboo Salt on Improvement of Helicobacter Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INSAN-HP-BS
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InSan Bamboo Salt (Experimental)
  Interventions: Dietary Supplement: InSan Bamboo Salt
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: InSan Bamboo Salt — InSan Bamboo Salt (10g/day)
  Arms: InSan Bamboo Salt
Dietary Supplement: Placebo — Placebo (10g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 4-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of InSan Bamboo Salt on improvement of Helicobacter pylori infection. The investigators measured improvement of Helicobacter pylori infection parameters , including 14C-UBT(Urea breath test), and subjects' symptoms, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-65 years old
* 14C-UBT test ≥ 100 cpm
* Endoscopy results showing gastritis
* Able to give informed consent

Exclusion Criteria:

* Diagnosed of gastrointestinal disease such as ulcer, cancer, more than 10 erosions
* Taken antibiotics and stomach medicines such as steroid, bismuth compound, H2-receptor antagonist and proton pump inhibitor within 2 weeks
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2013-07-25 (Actual); Study Completion 2013-07-25 (Actual)

PRIMARY OUTCOMES:
Changes in 14C-UBT(Urea breath test) | 4 weeks
  14C-UBT(Urea breath test) was measured in study visit 1(0 week) and visit 3(4 week).

SECONDARY OUTCOMES:
Changes in subjects' symptoms | 4 weeks
  subjects' symptoms was measured in study visit 1(0 week) and visit 3(4 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea